CLINICAL TRIAL: NCT05161429
Title: BESTMED: Observational Evaluation of Second Line Therapy Medications in Diabetes
Acronym: BESTMED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Baylor College of Medicine (Other); Baylor Scott and White Research Institute (Unknown); The Cleveland Clinic (Other); HealthCore, Inc. (Industry); Humana Inc. (Industry); Massachusetts General Hospital (Other); Medical Outcomes Management (Unknown); University of Iowa (Other); Allina Health (Unknown); Intermountain Health Care, Inc. (Other); Marshfield Clinic (Unknown); Medical College of Wisconsin (Other); University of Missouri-Columbia (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Alexander Turchin, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2021P001171
Record Dates: First submitted 2021-11-23; First posted 2021-12-17 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- DPP4: Patients receiving second line diabetes treatment with dipeptidyl peptidase-4 inhibitors (DPP4) following metformin
  Interventions: Drug: DPP4
- GLP1-RA: Patients receiving second line diabetes treatment with glucagon-like peptide-1 receptor agonists (GLP1-RA) following metformin
  Interventions: Drug: GLP-1 receptor agonist
- Basal insulin: Patients receiving second line diabetes treatment with basal insulin following metformin
  Interventions: Drug: Basal Insulin
- SLGT2: Patients receiving second line diabetes treatment with sodium-glucose cotransporter-2 inhibitors (SLGT2) following metformin
  Interventions: Drug: SLGT2
- SU: Patients receiving second line diabetes treatment with sulfonylureas (SU) following metformin
  Interventions: Drug: SU

INTERVENTIONS:
Drug: DPP4 — Dipeptidyl peptidase-4 inhibitors (DPP4) including alogliptin, linagliptin, sitagliptin, and saxagliptin
  Groups: DPP4
Drug: GLP-1 receptor agonist — Glucagon-like peptide-1 receptor agonists (GLP1-RA) including dulaglutide, exenatide, liraglutide and semaglutide
  Groups: GLP1-RA
Drug: Basal Insulin — degludec, detemir, glargine and NPH
  Groups: Basal insulin
Drug: SLGT2 — Sodium-glucose cotransporter-2 inhibitors (SLGT2) including canagliflozin, dapagliflozin, empagliflozin, and ertugliflozin
  Groups: SLGT2
Drug: SU — Sulfonylurea (SU) including glimepiride, glipizide, and glyburide
  Groups: SU

SUMMARY:
An observational study of electronic patient data to compare diabetes medications and to determine which ones offer the best balance of risks and benefits.

DETAILED DESCRIPTION:
Type 2 diabetes is an increasingly common disease that affects more than 10 percent of adults in the United States. Multiple medications are available to treat this condition. However, many of these medications have never been directly compared against one another, which makes it unclear which medication is the best to use.

Investigators will use a large database of electronic patient data to compare diabetes medications to determine which ones offer the best balance of risks and benefits. This database will draw from several large healthcare institutions and health insurance companies that collectively pull from a patient population of over 130 million across all major regions of the United States. Investigators will study adults aged 30 or older who have type 2 diabetes and are at moderate risk of heart attacks and strokes, and who are starting a second diabetes medication (after metformin). Investigators will use clinical trial emulation, a cutting-edge statistical technique, to compare the following classes of diabetes medications: (1) DPP4 inhibitors (alogliptin, linagliptin, sitagliptin, or saxagliptin); (2) GLP1 receptor agonists (dulaglutide, exenatide, liraglutide, or semaglutide); (3) basal insulin (degludec, detemir, glargine, or NPH); (4) SGLT2 inhibitors (canagliflozin, dapagliflozin, empagliflozin, or ertugliflozin); and (5) sulfonylureas (glimepiride, glipizide, or glyburide).

To determine which diabetes medications provide the greatest benefit to patients, investigators will compare how much they reduce the risks of the following \conditions: (1) heart attack; (2) heart failure; (3) stroke; (4) kidney disease; (5) eye disease; and (6) liver disease. To allow patients with diabetes and their doctors to make fully informed decisions about which diabetes medication to take, investigators will also compare these medications' risks of the following possible side effects: (1) low blood sugar; (2) kidney infection; (3) severe skin infections in the genital area; (4) foot/leg amputations; (5) broken bones; (6) pancreatitis (i.e., severe inflammation of the pancreas); (7) pancreatic cancer; (8) thyroid cancer; and (9) death from causes other than heart attacks or strokes.

In order to minimize the risk of bias and confounding, the analysis will be conducted using causal inference techniques, by emulating a randomized clinical trial (including both intention-to-treat and per-protocol analyses), while incorporating rigorous data quality checks.

ELIGIBILITY:
Individuals meeting the following criteria between January 1, 2015 and December 31, 2021:

* Diabetes mellitus (DM) type II
* HbA1c of 7-11% within the past year
* Monotherapy with metformin for at least 3 months
* No prior non-metformin outpatient diabetes therapy
* Aged ≥30y
* At "moderate" risk of ASCVD

  * Men aged ≥35y and women aged ≥45y with no history* of stroke, myocardial infarction, revascularization, or heart failure hospitalization
  * Men aged 30-34 and women aged 30-44 with history* of hypertension, hyperlipidemia, retinopathy, kidney disease or neuropathy
* estimated glomerular filtration rate (eGFR) ≥ 45 ml/min/1.73m2 within the past 3 years
* Not pregnant at time 0
* No history* of institutionalization with a diagnosis of dementia, metastatic cancer, end stage lung disease, end stage liver disease, pancreatitis, medullary thyroid cancer or severe UTIs
* Engagement with the healthcare system: enrollment for at least 12 months and attendance of at least one outpatient encounter in the prior 12 months

(*) History will be derived from at least 12 months of EHR and claims prior to time zero and will use all available EHR and claims data between January 1, 2014 and time zero

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is adults aged 30 or older who have type 2 diabetes and are at moderate risk of Atherosclerotic Cardiovascular Disease (ASCVD), and who are starting a second diabetes medication (after metformin). Patients from collaborating institutions will be included in the analysis based on study population inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 550000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
4-point major adverse cardiac events (MACE) | Follow-up begins 30 days after enrollment and ends at the earliest of a) the first study outcome; b) study end or c) loss to follow-up. Maximum duration of follow-up will be 10.5 years.
  Includes: a) death from cardiovascular causes b) non-fatal myocardial infarction (MI) c) non-fatal stroke and d) hospitalization for heart failure (HF)
3-point major adverse cardiac events (MACE) | Follow-up begins 30 days after enrollment and ends at the earliest of a) the first study outcome; b) study end or c) loss to follow-up. Maximum duration of follow-up will be 10.5 years.
  Includes: a) death from cardiovascular causes as reported in the National Death Index b) non-fatal MI and c) non-fatal stroke

SECONDARY OUTCOMES:
Adverse outcomes | Follow-up begins 30 days after enrollment and ends at the earliest of a) the first study outcome; b) study end or c) loss to follow-up. Maximum duration of follow-up will be 10.5 years.
  Includes a) severe hypoglycemia b) severe urinary tract infection (UTI) c) Fournier's gangrene d) lower extremity amputation e) bone fracture f) diabetic ketoacidosis (DKA) g) pancreatitis h) pancreatic cancer i) medullary thyroid cancer j) non-cardiovascular death
Severe clinical outcomes | Follow-up begins 30 days after enrollment and ends at the earliest of a) the first study outcome; b) study end or c) loss to follow-up. Maximum duration of follow-up will be 10.5 years.
  Includes: a) hospitalization for >= 30 days with any of the primary or secondary outcome endpoints as the primary or admitting diagnosis b) ICU admission with any of the primary or secondary outcome endpoints as the primary or admitting diagnosis or c) death from any cause
Non-cardiovascular outcomes | Follow-up begins 30 days after enrollment and ends at the earliest of a) the first study outcome; b) study end or c) loss to follow-up. Maximum duration of follow-up will be 10.5 years.
  Includes a) nephropathy b) diabetic retinopathy requiring treatment c) non-alcoholic fatty liver disease (NAFLD) with advanced fibrosis / nonalcoholic steatohepatitis (NASH)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Turchin, MD, MS, Principal Investigator — Brigham and Women's Hospital
Locations (5):
- United States (5):
  - HealthCore, Inc., Wilmington, Delaware
  - Humana, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Greater Plains Collaborative, Beachwood, Ohio
  - Baylor Scott & White, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson PW, D'Agostino RB, Levy D, Belanger AM, Silbershatz H, Kannel WB. Prediction of coronary heart disease using risk factor categories. Circulation. 1998 May 12;97(18):1837-47. doi: 10.1161/01.cir.97.18.1837. PMID 9603539
- [Background] D'Agostino RB, Wolf PA, Belanger AJ, Kannel WB. Stroke risk profile: adjustment for antihypertensive medication. The Framingham Study. Stroke. 1994 Jan;25(1):40-3. doi: 10.1161/01.str.25.1.40. PMID 8266381
- [Background] Kannel WB, D'Agostino RB, Silbershatz H, Belanger AJ, Wilson PW, Levy D. Profile for estimating risk of heart failure. Arch Intern Med. 1999 Jun 14;159(11):1197-204. doi: 10.1001/archinte.159.11.1197. PMID 10371227